CLINICAL TRIAL: NCT00515047
Title: Genetics of Atopic Dermatitis - Eczema Herpeticum
Brief Title: Identifying Genetic Determinants of Eczema Herpeticum and Other Viral Infections in Individuals With Atopic Dermatitis
Acronym: Genetics
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ADVN GENE 04; HHSN266200400033
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema; Eczema Herpeticum; Molluscum Contagiousum; Herpes Simplex; Vaccinia
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Kaposi Varicelliform Eruption; Herpes Simplex; Vaccinia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin scrapings and blood collection may occur
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Eczema Herpeticum (EH): Participants with AD who currently have or have had EH
- Non-EH: Participants with AD who do not have and have never had EH
- Healthy Controls: Healthy participants without a history of AD

SUMMARY:
People with atopic dermatitis (AD), or eczema, are susceptible to skin infections and inflammations. Some individuals with AD develop a condition known as eczema herpeticum (EH) following exposure to the herpes simplex virus (HSV). The purpose of this study is to identify the genetic determinants that lead people with AD to develop EH and similar conditions caused by other viruses.

DETAILED DESCRIPTION:
AD is a chronic inflammatory skin disorder characterized by recurrent viral skin infections. However, people with AD do not all develop the same infections. For example, some people with AD who receive the smallpox vaccine develop a life-threatening condition known as eczema vaccinatum (EV). This study focuses on individuals with AD who also have a history of eczema herpeticum (ADEH+), a condition similar to EV. It is unlikely that the differences in the development of skin infections are due to differences in viral exposure, and instead due to differences in each individual's response to viruses. The purpose of this study is to determine the genetic pathways which are responsible for the development of viral skin infections in people with AD.

Participants in this study will also be enrolled in the ADVN Biomarker Registry Study. There will be only one clinical visit for this study at which blood and/or skin samples may be collected. The samples will then have high-throughput genotyping to define genetic markers in individuals susceptible to viral infections.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in ADVN Biomarker Registry Study
* Non-Hispanic and only African American or only Caucasian race
* Parent or guardian willing to provide informed consent, if necessary

Exclusion Criteria:

* History of any systemic illness, excluding AD
* Participation of a first degree relative already enrolled in the genotyping study unless the subject in question fulfills the diagnostic criteria for ADEH+. More information on this criterion can be found in the protocol.

Ages: 8 Months to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: African-American, Caucasian, and Non-Hispanic people ages 8 months to 80 years
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2006-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Identification of variants/haplotypes in EH-associated genes and characterization of frequencies of variants in priority candidate genes for EH | Throughout Study

SECONDARY OUTCOMES:
Identification and prioritization of novel genes induced in response to viral infection (HSV/Vaccinia and MCV) in AD participants and relevant control groups | Throughout Study

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beck, MD, Principal Investigator — University of Rochester; Kathleen Barnes, PhD, Principal Investigator — Johns Hopkins Allergy and Asthma Center
Locations (7):
- United States (7):
  - University of California at San Diego, La Jolla, California
  - National Jewish Health, Denver, Colorado
  - Children's Memorial Hospital, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Oregon Health & Sciences University, Portland, Oregon

REFERENCES:
- [Background] Baker BS. The role of microorganisms in atopic dermatitis. Clin Exp Immunol. 2006 Apr;144(1):1-9. doi: 10.1111/j.1365-2249.2005.02980.x. PMID 16542358
- [Background] Kim BE, Leung DY, Streib JE, Kisich K, Boguniewicz M, Hamid QA, Howell MD. Macrophage inflammatory protein 3alpha deficiency in atopic dermatitis skin and role in innate immune response to vaccinia virus. J Allergy Clin Immunol. 2007 Feb;119(2):457-63. doi: 10.1016/j.jaci.2006.10.005. Epub 2006 Dec 4. PMID 17141855
- [Background] Porter CD, Muhlemann MF, Cream JJ, Archard LC. Molluscum contagiosum: characterization of viral DNA and clinical features. Epidemiol Infect. 1987 Oct;99(2):563-6. doi: 10.1017/s0950268800068072. PMID 2824227
- [Background] Umene K, Yoshida M, Sakaoka H. Comparison of the association with eczema herpeticum in the two predominant genotypes of herpes simplex virus type 1. J Med Virol. 1996 Aug;49(4):329-32. doi: 10.1002/(SICI)1096-9071(199608)49:43.0.CO;2-5. PMID 8877767
- [Result] Gao PS, Leung DY, Rafaels NM, Boguniewicz M, Hand T, Gao L, Hata TR, Schneider LC, Hanifin JM, Beaty TH, Beck LA, Weinberg A, Barnes KC. Genetic variants in interferon regulatory factor 2 (IRF2) are associated with atopic dermatitis and eczema herpeticum. J Invest Dermatol. 2012 Mar;132(3 Pt 1):650-7. doi: 10.1038/jid.2011.374. Epub 2011 Nov 24. PMID 22113474
- [Result] Gao PS, Rafaels NM, Mu D, Hand T, Murray T, Boguniewicz M, Hata T, Schneider L, Hanifin JM, Gallo RL, Gao L, Beaty TH, Beck LA, Leung DY, Barnes KC. Genetic variants in thymic stromal lymphopoietin are associated with atopic dermatitis and eczema herpeticum. J Allergy Clin Immunol. 2010 Jun;125(6):1403-1407.e4. doi: 10.1016/j.jaci.2010.03.016. Epub 2010 May 13. No abstract available. PMID 20466416
- See also: Click here for more information about the Atopic Dermatitis and Vaccinia Network — http://www.nationaljewish.org/adrn/index/